CLINICAL TRIAL: NCT00876278
Title: Prospective Clinical Study to Evaluate Usability of Mesotest II for Assessment of Night Driving Capacity of Pseudophakic Patients Implanted With Monofocal IOL *AT.Smart 46LC
Brief Title: Night Driving Pilot
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to internal reasons study was not performed.
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 46LC HEN 401-08
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Cataract
Keywords: Cataract; Intraocular Lens (IOL); Mesotest II; Evaluation of usability of Mesotest II for assessment of night driving capacity of pseudo-phakic patients
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- *AT.Smart 46LC (Other): The *AT.Smart 46LC is indicated for primary implantation for the visual correction of aphakia in persons in whom the cataractous lens has been removed by phacoemulsification extracapsular cataract extraction. The IOL is intended to be placed only in an intact capsular bag. When implanted, the *AT.Smart 46LC replaces the natural lens of the eye and functions as a refracting medium in the correction of aphakia.
  Interventions: Device: *AT.Smart 46LC

INTERVENTIONS:
Device: *AT.Smart 46LC — Primary implantation of *AT.Smart 46 LC into the eye's capsular bag for the visual correction of aphakia in persons in whom the cataractous lens has been removed by phacoemulsification extracapsular cataract extraction. The IOL is intended to be placed only in an intact capsular bag. When implanted, the *AT.Smart 46LC replaces the natural lens of the eye and functions as a refracting medium in the correction of aphakia.

SUMMARY:
Pilot study to evaluate usability of Mesotest II for assessment of night driving capacity of pseudo-phakic patients implanted with aspheric monofocal posterior chamber IOL *AT.Smart 46LC.

Target Criterion:

Measurement of contrast sensitivity and sensitivity to light under mesopic conditions (Mesotest II, Oculus).

ELIGIBILITY:
Inclusion Criteria:

* Healthy eyes with cataract
* Patient age 50-75 years
* Written Patient Informed Consent
* Assured follow-up examination

Exclusion Criteria:

* Any kind of macula degeneration and impairment of retina (clinical diagnosis)
* Amblyopia
* Intraoperative complications; damaged posterior bag; intraocular haemorrhage
* Astigmatism > 1.5 D (objective, preoperative)
* Pregnancy or lactation period for female patients

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of contrast sensitivity and sensitivity to light under mesopic conditions (Mesotest II, Oculus). | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J. Mueller, MD, Principal Investigator — Klinikum Augsburg, Klinik für Augenheilkunde
Locations (1):
- Klinikum Augsburg, Klinik für Augenheilkunde, Augsburg, Germany